CLINICAL TRIAL: NCT01705912
Title: Fall Prevention by Assistant Nurses Among Community Living Elderly With Risk of Falling - a Randomized Controlled Trial
Brief Title: Fall Prevention Among Community Living Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gunilla Fahlstrom (Other Government)
Collaborators: Örebro County Council (Other Government); Örebro University, Sweden (Other)
Responsible Party: Sponsor-Investigator, Gunilla Fahlstrom, PhD, Örebro County Council
Organization: Örebro County Council (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OLLGF01; OLLGF0112 (Other: Orebro county council)
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Accidental Falls/Prevention and Control
Keywords: fall; prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Experimental): Complete intervention i.e. basic intervention + individual training program.
  Interventions: Other: Complete intervention
- Control (Active Comparator): Basic intervention.
  Interventions: Other: Basic intervention

INTERVENTIONS:
Other: Complete intervention — The basic intervention, an occupational therapist assessed the home environment and gave advice, if necessary. Then participants were assessed by a physiotherapist concerning health and function pre and post intervention. The intervention consisted of an individually designed home exercise program aiming at improving balance, muscle strength and walking ability. The program, which was made by the physiotherapist, should be performed three times a week. A minimum of 30 minutes of walking per week was recommended, encouring further walking on an individual basis. An assistant nurse made eight home visits to supervise, help and encourage performance of activities.
  Arms: Training
Other: Basic intervention — The basic interventions was an occupational therapist assessed the home environment and gave advice, if necessary. Then participants were assessed by a physiotherapist concerning health and function pre and post intervention.
  Arms: Control

SUMMARY:
The purpose of this study is to assess effects of a home exercise program, supervised by assistant nurses with the aim of preventing falls.

Community living persons 65 years of age or older having a risk of falling were invited to participate. Participants were randomized to either training or control.

The training program was individually designed by a physiotherapist and the 5-month program performance was supervised in the partcipants home by eight home visits from an assistant nurse.

All participants received a visit from an occupational therapist who assessed the home and, if necessary, gave advice.

DETAILED DESCRIPTION:
Falls among elderly are a major public health problem, but preventive interventions containing physical exercise and home improvement are available.

In this study the crucial question was to test whether unlicensed staff, assistant nurses, could be used for preventive work.

Estimation of study power gave that 170 participants in each group would be needed to detect a difference in days with falls, the main outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* community living persons at least 65 years old
* independent walking ability with or without walking aid
* experienced at least one fall during the last 12 months
* ability to communicate and cooperate with study staff

Exclusion Criteria:

* ongoing physiotherapy treatment
* ongoing participation in exercise/acitivity containing balance and strength enhancing components
* a dementia diagnose
* mental disorder that affects possibility to communicate and cooperate
* other medical reason making participation inte the study inappropriate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 148 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of days with fall | 12 months
  Self reported calendar data

SECONDARY OUTCOMES:
Exercise | 12 months
  Self reported calendar data

OTHER OUTCOMES:
Strength | Pre and post intervention, 5 months
  Chair stand test
Balance | Pre and post intervention, 5 months
  Falls efficacy scale (FES)
Balance | Pre and post intervention, 5 months
  Bergs balance scale
Walking 3 metres test | Pre and post intervention, 5 months
Health related quality of life | Pre and post intervention, 5 months
  Self reported interview data, SF-36
Activities of daily living | Pre and post intervention, 5 months
  ADL
Walking | 12 months
  Minutes of walking per day, self reported calendar data.
Hospital days | 12 months
  Hospital register data
Hospital visits | 12 months
  Hospital register data
Fractures or other harms | 12 months
  Hospital register data
Strength | Pre and post assessment, 5 months
  Timed Up and Go, TUG

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Fahlstrom, PhD, Principal Investigator — Örebro County Council
Locations (1):
- Family medicine research center, Örebro, Sweden